CLINICAL TRIAL: NCT03944629
Title: Efficacy of Arnica Montana in Reducing Postoperative Edema and Pain Following Third Molar Extraction
Brief Title: Efficacy of Arnica Montana in Reducing Postoperative Edema and Pain
Status: Completed | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12692
Record Dates: First submitted 2018-02-15; First posted 2019-05-09 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Arnica; Third Molar Extraction
MeSH Terms: interventions — Arnicae flos extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: To decrease bias, this study will be double blinded by blinding information about the specific group from the subject and the investigators. The study medication and matching placebo (sugar pill) will be blinded and packaged in blister cards provided by the Sponsor.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Study Group (Experimental): The study group will be comprised of subjects who will receive homeopathic Arnica montana (SinEcch™) for perioperative management of edema and pain.
  Interventions: Drug: SinEcch
- Control Group (Placebo Comparator): The control group will be comprised of subjects who will receive matching SinEcch™ placebo (sugar pill).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SinEcch — The study group will be comprised of subjects who will receive homeopathic Arnica montana (SinEcch™) for perioperative management of edema and pain.
  Other Names: Arnica montana
  Arms: Study Group
Other: Placebo — The control group will be comprised of subjects who will receive matching SinEcch™ placebo (sugar pill).
  Arms: Control Group

SUMMARY:
This study is a prospective, randomized, double-blinded, controlled, clinical trial that evaluates the efficacy of using high potency homeopathic Arnica montana (SinEcch™) during the perioperative period for decreasing swelling and pain after extraction of partial or full/complete bony impacted third molars. The study group will be comprised of subjects who will receive homeopathic Arnica montana (SinEcch™) for perioperative management of edema and pain. The control group will be comprised of subjects who will receive matching SinEcch™ placebo (sugar pill).

DETAILED DESCRIPTION:
Our study aims to look at the efficacy of homeopathic Arnica montana (SinEcch™) in reducing postoperative edema and pain. Pain will be measured using the visual analog scale (VAS). Swelling will be measured using a 3D imaging system. This is the first study using the 3D imaging system that looks at the effect of homeopathic Arnica montana in reducing facial swelling following the surgical removal of impacted third molars. Although SinEcch is marketed mainly for management of postoperative swelling and bruising, Arnica Montana has been used for managing the sequelae of postoperative inflammation including pain so one of the secondary outcome measure for this study is to measure the efficacy of SinEcch in management of post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex and of any race from the ages of 18 to 40 years.
* Subjects for whom a decision has been made to extract 4 third molars, and who have at least 2 of third molar teeth classified as full or partially bony impacted in the mandible, and they will be evaluated to have at least 2 of third molar teeth classified as erupted or impacted (full or partially bony) in the maxilla under local anesthesia alone, local anesthesia and sedation, or local anesthesia and general anesthesia, all in an outpatient setting.

  1. Full/complete bony: The entire tooth is below the level of the alveolar bone. The tooth is completely encased in bone so that when the gingiva is cut and reflected back, the tooth is not seen. Bone removal (large amounts) together with root sectioning will be needed to remove the tooth.
  2. Partial bony: A portion of the height of the contour of the tooth is below the level of the alveolar bone. The superficial portion of the tooth is covered only by soft tissue, but the height of the tooth's contour is below the level of the surrounding alveolar bone.
* Subjects must be physically able to tolerate conventional surgical procedures (ASA I/II).
* Subjects must agree to follow the study protocol as shown by signing the informed consent form.

Exclusion Criteria:

* Subjects who are known to be pregnant or think they may be pregnant. (A urine pregnancy test will be performed on female subjects at Day 0 - Visit 1. Subjects testing positive will be excluded from study participation.)
* Subjects with skeletal immaturity as determined by the medical history.
* Subjects with self-reported current or history of substance abuse.
* Subjects who are currently receiving any anti-inflammatory or pain medication chronically, or they suffer from a chronic pain condition.
* Subjects with an allergy to Vicodin (or its constituents, acetaminophen and hydrocodone).
* Subjects who are diagnosed with fibromyalgia.
* Allergy to ragweed and other related plants.
* Subjects with an allergy to hypromellose.
* Non-English speaking patients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine Department of Oral and Maxillofacial Surgery, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 27 | 26
Completed | 26 | 24
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 22.4 [18 to 28] | 23.5 [18 to 36] | 22.95 [18 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 12 | 13 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 6 | 15
  African American | 3 | 3 | 6
  White | 9 | 11 | 20
  Hispanic/Latino | 3 | 3 | 6
  Multi | 2 | 2 | 4
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53
BASELINE Postoperative Swelling [Mean (Standard Deviation); unit: Cm^2]
  Right Side | 40.6264 (23.21150) | 45.9915 (27.64742) | 43.30895 (2.68255)
  Left Side | 40.589 (23.28939) | 45.0376 (23.79449) | 42.8133 (2.2243)
BASELINE PAIN [Mean (Standard Deviation); unit: units on a scale] — This represents pain that the participant would indicate, through units on a scale, as a way to reflect the level of pain they are in immediately following their surgery, before any study intervention begins.
  units on a scale | 0.4259 (1.53788) | 0.2712 (0.80302) | 0.34855 (0.07735)

OUTCOME MEASURES:

1. Primary Outcome: Change in Postoperative Facial Swelling From Baseline to Day 3
Description: Primary outcome is the change in postoperative facial swelling volume as measured by the 3dMD™ system
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 27 | 26
cm^2
  Right Side | 9.2508 (10.29876) | 9.3320 (13.95499)
  Left Side | 7.4336 (9.57758) | 7.0346 (12.41098)

2. Primary Outcome: Change in Postoperative Facial Swelling From Day 3 to Day 5
Description: Primary outcome is the change in postoperative facial swelling volume as measured by the 3dMD™ system
Time Frame: Day 3 and Day 5
Population: three subjects did not complete the day 5 visit and thus, data was only analyzed for 50 subjects instead of 53.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 26 | 24
cm^2
  Right Side | -1.9433 (8.22751) | -1.7292 (9.08343)
  Left Side | -3.225 (8.90529) | -2.6692 (10.96405)

3. Primary Outcome: Change in Postoperative Facial Swelling From Baseline to Day 5
Description: Primary outcome is the change in postoperative facial swelling volume as measured by the 3dMD™ system
Time Frame: Baseline and Day 5
Population: three subjects did not complete the day 5 visit and thus, data was only analyzed for 50 subjects instead of 53.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 26 | 24
cm^2
  Right Side | 7.6311 (7.76589) | 5.7718 (12.17906)
  Left Side | 4.4662 (10.41910) | 2.7803 (12.07358)

4. Secondary Outcome: Change in Post Operative Pain From Baseline to Day 3
Description: Change in postoperative pain as measured by 0-100 mm Visual Analog Scale, from baseline to post-operative Day 3, and from baseline to post-operative Day 5 (0 being the least pain, 100 being the most pain)
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 27 | 26
score on a scale | 1.741 (1.889) | 2.248 (1.98)

5. Secondary Outcome: Change in Post Operative Pain From Baseline to Day 5
Description: as for outcome 4
Time Frame: Baseline and Day 5
Population: three subjects did not complete the day 5 visit and thus, data was only analyzed for 50 subjects instead of 53.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 26 | 24
score on a scale | 0.523 (1.186) | 0.935 (1.077)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03944629/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03944629/ICF_004.pdf